CLINICAL TRIAL: NCT07374627
Title: Vertical Root Extraction for Immediate Implant Placement : A Prospective Clinical And Radiographic Single Arm Study.
Brief Title: Vertical Root Extraction for Immediate Implant
Acronym: Benex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mihad Ibrahim, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-056
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Implant Placement in Maxillary Esthetic Zone; Immediate Dental Implant Loading
Keywords: Dental Implant; root extraction

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, randomized, two-arm, parallel assignment clinical trial with a 1:1 allocation ratio. Eligible participants with a single hopeless maxillary anterior tooth indicated for extraction will be randomly assigned to one of two groups:
  Test Group (Benex Vertical Extraction): Patients will undergo flapless vertical root extraction using the Benex system, followed immediately by implant placement using a standardized guided protocol.
  Control Group (Conventional Atraumatic Extraction): Patients will undergo atraumatic incisal extraction with periotomes and forceps, followed immediately by implant placement using the same implant system and surgical protocol.
  Both groups will follow identical implant placement, grafting (if needed), provisionalization, and restoration procedures. The only variable between the groups is the extraction technique. Randomization will be computer-generated and concealed in sealed opaque envelopes. Surgeons cannot be blinded due
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benex (Experimental): Participants in this arm will undergo flapless vertical root extraction using the Benex system, followed immediately by implant placement with a standardized guided surgical protocol. The Benex system applies controlled vertical traction through a screw anchored in the root canal, minimizing lateral forces and reducing trauma to the socket walls. All patients will receive the same implant system, grafting material if indicated, provisional restoration, and final prosthesis according to the study protocol.
  Interventions: Procedure: vertical extraction
- Control (Active Comparator): Participants in this arm will undergo atraumatic incisal extraction using periotomes and forceps, followed immediately by implant placement with the same implant system and surgical protocol as the test group. This represents the current conventional method of atraumatic extraction. All subsequent implant placement, grafting (if needed), provisionalization, and final restoration steps will be standardized and identical to the test group.
  Interventions: Procedure: Conventional exctraction

INTERVENTIONS:
Procedure: vertical extraction — Participants in this arm will undergo flapless vertical root extraction using the Benex system, followed immediately by implant placement with a standardized guided surgical protocol. The Benex system applies controlled vertical traction through a screw anchored in the root canal, minimizing lateral forces and reducing trauma to the socket walls. All patients will receive the same implant system, grafting material if indicated, provisional restoration, and final prosthesis according to the study protocol.
  Arms: Benex
Procedure: Conventional exctraction — Tooth extraction is one of the most common procedures in dentistry, forming a cornerstone of both general dental practice and surgical specialties such as oral surgery and periodontology. Traditional extraction methods often involved the use of elevators and forceps to apply significant lateral and rotational forces, which could traumatize the alveolar bone and soft tissues. Over the past few decades, with the rise of implant dentistry and the need to preserve bone for future prosthetic rehabilitation, clinicians have shifted towards atraumatic extraction techniques. These methods aim to remove teeth while minimizing damage to surrounding hard and soft tissues, particularly the delicate alveolar socket walls.
  Arms: Control

SUMMARY:
Immediate implant placement in the esthetic zone has become a preferred treatment modality due to its potential to shorten treatment duration, reduce surgical interventions, and preserve the natural contour of peri-implant tissues (Chen & Buser, 2009; Lang et al., 2012). Despite these advantages, the technique remains surgically demanding, especially in the anterior maxilla, where the labial plate is often thin and highly susceptible to post-extraction resorption (Spray et al., 2000; Chappuis et al., 2017).

The greatest dimensional changes in alveolar ridge volume occur within the first 8-12 weeks after tooth extraction, with reductions in both height and width of the buccal bone crest (Araújo & Lindhe, 2005; Tan et al., 2012). This remodeling compromises mucogingival architecture, often leading to mid-facial soft tissue recession and esthetic failures. Conventional extraction methods, which apply rotational or lateral forces using elevators and forceps, risk fracturing the socket walls and accelerating bone loss (Araujo & Lindhe, 2009; Oghli & Steveling, 2010).

The introduction of atraumatic extraction systems aimed to address this challenge. The Benex vertical extraction system operates by inserting a screw into the root canal and applying controlled vertical traction. This approach minimizes lateral stress on socket walls, theoretically preserving the thin labial plate, which is critical for esthetic success (Muska et al., 2013; Canellas et al., 2021). Vertical traction avoids socket expansion and microfractures, enabling safer immediate implant placement in compromised situations.

Case reports and retrospective series have demonstrated encouraging clinical results with Benex, including intact labial plates on CBCT, high implant survival, and favorable Pink Esthetic Scores (Fürhauser et al., 2005; Canellas et al., 2021). Patients also report reduced discomfort and trauma perception, suggesting potential psychosocial benefits. However, most of the current evidence is based on small-scale case series (Blus & Szmukler-Moncler, 2010; Singla & Sharma, 2020), and randomized controlled trials comparing Benex-assisted extraction with conventional atraumatic extraction are lacking.

A robust RCT evaluating both objective esthetic outcomes (Midfacial mucosal recession, PES, CBCT bone preservation) and subjective patient-reported outcomes (PROMs) is therefore essential to validate the clinical value of the Benex system in the esthetic zone.

DETAILED DESCRIPTION:
The esthetic zone poses unique challenges for immediate implant placement due to the delicate nature of the labial bone. Several systematic reviews have shown that the thickness of the facial bone strongly influences marginal bone loss and soft tissue stability (Spray et al., 2000; Chappuis et al., 2017). Thin buccal plates (<1 mm) are particularly prone to resorption, with poor prognosis for soft tissue esthetics if damaged during extraction.

Ridge alterations after extraction. Araújo & Lindhe (2005) in an experimental model, and Tan et al. (2012) in humans, confirmed substantial horizontal and vertical resorption within weeks of extraction, with the labial wall showing the greatest reduction. Botticelli et al. (2004) and Iasella et al. (2003) demonstrated that ridge preservation measures reduce, but do not eliminate, resorption.

Atraumatic extraction techniques. Conventional methods using forceps and elevators often damage interproximal and buccal bone (Araujo & Lindhe, 2009). To counter this, atraumatic extraction devices were developed, such as periotomes (Sharma et al., 2015), piezosurgery (Blus & Szmukler-Moncler, 2010), and vertical extraction systems like Benex, Physics Forceps, and Sapian kits (Muska et al., 2013; Jain & Sridevi, 2016). These techniques reduce trauma and facilitate immediate implant placement, though operator skill and case selection remain crucial.

Benex system evidence. Muska et al. (2013) provided proof-of-principle for vertical extraction, showing intact socket walls and reduced risk of root fracture compared to forceps. Case series using Benex reported intact labial plates and favorable implant outcomes, but highlighted limitations in multirooted teeth and endodontically treated roots (Hong et al., 2018). Canellas et al. (2021) systematically reviewed atraumatic extractions, concluding that while vertical extraction devices appear promising, evidence is limited and heterogeneous.

Pink Esthetic Score (PES). Introduced by Fürhauser et al. (2005), the PES provides a standardized evaluation of peri-implant esthetics, including papillae, soft tissue level, contour, and color. PES has become the benchmark for clinical trials assessing esthetic outcomes of immediate implant protocols. High PES scores are closely linked to intact labial plates and preserved soft tissue contours (Chappuis et al., 2017).

Recent clinical trials. Ghallab et al. (2022) conducted a randomized controlled trial comparing vestibular and incisal extraction techniques within a vestibular socket therapy protocol. The vestibular approach demonstrated superior soft tissue stability and higher PES compared to incisal extraction. This supports the hypothesis that the extraction method critically determines esthetic outcomes. However, RCTs specifically testing vertical extraction systems like Benex are absent.

Knowledge gap. Current evidence suggests that vertical extraction systems may preserve bone and soft tissue better than conventional atraumatic methods. Yet, without randomized trials, their true clinical value remains uncertain. This trial aims to fill that gap by systematically evaluating Benex-assisted extraction versus conventional atraumatic extraction, focusing on both radiographic and patient-reported outcomes at 6 months.

ELIGIBILITY:
Inclusion Criteria:

- dults aged 18 to 55 years. Classified as ASA I-II (healthy or mild systemic condition, fit for surgery). The presence of a single hopeless maxillary anterior tooth (incisor or canine) indicated for extraction.

Adequate palatal and apical bone volume to achieve primary stability for immediate implant placement.

Patients are able and willing to provide informed consent and comply with study visits.

Exclusion Criteria:

Smokers consuming more than 10 cigarettes per day. Pregnant or lactating women. Patients with systemic contraindications to surgery (e.g., chemotherapy, radiotherapy, bisphosphonate therapy).

Patients with untreated periodontal disease. Presence of active local infection at the surgical site.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mid facial recession | 6 months
  The vertical change in the soft tissue margin at the mid-facial aspect of the implant crown compared to baseline (immediately after provisionalization). This will be measured in millimeters using standardized calibrated intraoral photographs. Positive values indicate soft tissue recession, and negative values indicate coronal migration.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Shalash, Study Director — National Research Centre, Egypt
Locations (1):
- Cairo University, Cairo, Egypt